CLINICAL TRIAL: NCT03918395
Title: Does Protein and Polyphenol Supplementation Augment Adaptations to 30 Sessions of Resistance Exercise Training in Healthy Males and Females Compared to an Isoenergetic Placebo Supplement?
Brief Title: Supplemental Protein And Resistance Training Adaptations
Acronym: SPARTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 171206/B/09
Record Dates: First submitted 2019-04-16; First posted 2019-04-17 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Hypertrophy
MeSH Terms: conditions — Hypertrophy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo beverage
  Interventions: Dietary Supplement: Placebo beverage
- Protein-Polyphenol supplement (Active Comparator): Protein-polyphenol beverage
  Interventions: Dietary Supplement: Protein-polyphenol beverage

INTERVENTIONS:
Dietary Supplement: Placebo beverage — A placebo beverage will be consumed both post-exercise and pre-bed
  Arms: Placebo
Dietary Supplement: Protein-polyphenol beverage — A protein-polyphenol beverage will be consumed both post-exercise and pre-bed
  Arms: Protein-Polyphenol supplement

SUMMARY:
Chronic resistance training has been shown to increase muscle cross-sectional area, volume and strength. Individuals participating in a resistance training program may wish to consume protein supplements to aid recovery and maximise adaptation. Furthermore, antioxidants have been shown to aid recovery from acute bouts of exercise. However, the effect of antioxidants combined with protein on long term-training adaptation is not fully understood.

This study will combine measures of muscle size, muscle strength and function, and the underlying changes in muscle metabolism in order to assess the effect of consuming a combined protein-antioxidant supplement during a 30 session resistance training program.

DETAILED DESCRIPTION:
Supplemental protein ingestion is an established method for augmenting gains in fat free mass, muscle strength and muscle cross sectional area following a period of resistance exercise training. In addition to protein, supplements high in polyphenols such as berry and pomegranate extract are believed to be an effective method of reducing soreness and facilitating recovery following a single bout of resistance exercise.

However, whilst polyphenols are shown to facilitate recovery from a single session of resistance exercise, their effect on adaptations to repeated bouts of resistance exercise are unknown. Asking this question will allow a detailed investigation of the mechanisms by which protein-polyphenol ingestion may affect adaptations to resistance exercise training when compared to a non protein or polyphenol containing placebo, which is an important yet underexplored area

ELIGIBILITY:
Inclusion Criteria:

* Male and Female
* 18 - 40 years of age
* Recreationally active

Exclusion Criteria:

* Any diagnosed metabolic impairment (e.g. type 1 or 2 Diabetes). Such impairments can affect skeletal muscle metabolism
* Any diagnosed cardiovascular disease or hypertension
* Use of nutritional supplements (e.g. protein, polyphenols, vitamins, antioxidants) as use of nutritional supplements during the study period may interfere with the physiological responses to the supplements of interest administered in this study.
* Habitual dietary protein intake <0.8 g/kg/day or >1.6 g/kg/day as calculated with a three day diet diary. Habitually low protein may impair adaptations to resistance exercise training and a habitually excessive protein intake may negate the benefit of protein supplementation.
* Current musculoskeletal injury that may impair exercise performance or may be exacerbated due to this studies exercise protocol.
* Resistance trained (participating in structured resistance exercise 3 or more times per week for >6 months), endurance trained (participating in structured endurance exercise for >6h per week for >6 months), or sedentary participants as these are not the populations of interest.
* Chronic use of anti-inflammatory medicines prior to the study and unwillingness to refrain from taking anti-inflammatory medications during the study as these medications may affect skeletal muscle metabolism and/or adaptation to exercise.
* Individuals who carry an epi-pen, or those with a diagnosed allergy or who believe that they have an allergy to milk or milk products, crustacean shellfish, tree nuts, or peanuts
* Individuals with a severe allergy to egg, fish, wheat or soy ingredients as the product is manufactured in a facility that contains these ingredients
* Individuals with non removable metallic implants (including heart pacemaker, cochlea implants, medication pumps, surgical clips, plates or screws) or claustrophobia

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-12-21 (Actual); Study Completion 2019-12-21 (Actual)

PRIMARY OUTCOMES:
Change in cross-sectional area of quadriceps muscle group | After 30 training sessions (approx. 10 weeks)
  The cross-sectional area of the muscles comprising the thigh after 30 training sessions will be compared to pre-training values. This will be measured using MRI.

SECONDARY OUTCOMES:
Change in quadriceps muscle group volume | After 30 training sessions (approx. 10 weeks)
  The volume of the muscles comprising the thigh after 30 training sessions will be compared to pre-training values. This will be measured using MRI.
Change in knee extensor isokinetic total work | After 30 training sessions (approx. 10 weeks)
  Bilateral knee extensor isokinetic total work will be assessed before and after the training program by quantifying work completed over 30 isokinetic quadriceps contractions on an isokinetic dynamometer.
Change in maximal isometric peak torque | After 30 training sessions (approx. 10 weeks)
  Knee extensor isometric peak torque will be assessed before and after the training program using an isokinetic dynamometer.
Change in maximal isokinetic peak torque | After 30 training sessions (approx. 10 weeks)
  Knee extensor isokinetic peak torque over 3 repetitions will be assessed before and after the training program using an isokinetic dynamometer.
Change in muscle protein synthesis assessed using the stable isotope Deuterium Oxide | After 30 training sessions (approx. 10 weeks)
  The enrichment of deuterated alanine (from the deuterium oxide heavy water stable isotope tracer) in vastus lateralis biopsy samples will be measured relative to the non-deuterated alanine. The change over 48 hours will be measured pre- and post-training to calculate a fractional synthesis rate (% day).
Perceived quadriceps muscle soreness: | After 30 training sessions (approx. 10 weeks)
  Soreness will be assessed at the start of each training session using a validated visual analogue scale (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Francis Stephens, PhD, Principal Investigator — University of Exeter
Locations (1):
- University of Exeter, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No